CLINICAL TRIAL: NCT02748304
Title: A Prospective Randomized Control Trial of the Effect of Sorafenib Combined With Aspirin in Preventing the Recurrence in High-risk Patients With Hepatocellular Carcinoma
Brief Title: Sorafenib Combined With Aspirin to Prevent the Recurrence in High-risk Patients With Hepatocellular Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The enrollment of this study was slow. With the approval of lenvatinib in HCC,many patients choose the new drug, so subsequent enrollment may be more difficult.
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lunxiu Qin, Director of the general surgery department, Huashan hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Huashan 003
Record Dates: First submitted 2016-04-12; First posted 2016-04-22 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Aspirin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (Placebo Comparator): just follow up after liver resection in HCC patients
  Interventions: Other: control
- sorafenib (Active Comparator): use sorafenib after liver resection in HCC patients
  Interventions: Drug: sorafenib
- sorafenib and aspirin (Active Comparator): use sorafenib and aspirin after liver resection in HCC patients
  Interventions: Drug: sorafenib; Drug: aspirin

INTERVENTIONS:
Other: control — just follow up
  Arms: control
Drug: sorafenib — sorafenib 400mg bid po
  Other Names: sorafenib treatment
  Arms: sorafenib; sorafenib and aspirin
Drug: aspirin — aspirin 100mg qd po
  Other Names: aspirin treatment
  Arms: sorafenib and aspirin

SUMMARY:
The purpose of the study is to observe the effect of sorafenib combined with aspirin in preventing the recurrence in high-risk patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
The recurrence of hepatocellular carcinoma(HCC）is the main problem during the treatment. Although some methods such as interferon may be effective in preventing the recurrence, there is still no clear effective approach widely accepted for everyone.

Sorafenib, a kind of tyrosine kinase inhibitor, which inhibiting proliferation and inducing apoptosis of tumor cell by inhibiting the raf/MEK/ERK pathway, and anti-angiogenesis by targeting Vascular Endothelial Growth Factor Receptor(VEGFR), has now become the standard treatment of advanced HCC patients. Although the STORM studies have shown that adjuvant sorafenib for such patients did not significantly affect recurrence-free survival, time to recurrence, or overall survival. The patients recruiting in the study were mostly early stage, for middle and late stage patients, whether sorafenib can reduce tumor recurrence after surgical resection and prolong survival remains to be further study.

Aspirin is a kind of nonsteroidal anti-inflammatory drugs. It is the first hint of aspirin's potential role in tumor prevention and treatment when Gasic found that tumor metastasis is reduced in thrombocytopenia mice, and then the research confirmed that aspirin treatment can significantly reduce the tumor metastasis. In recent years, a lot of epidemiological evidence and clinical trials found that aspirin played an important role in cancer prevention, at the same time, more experimental study has found that it can also play a role in tumor treatment. Our previous animal experiments found that a combination of sorafenib and aspirin can reverse the negative effect of sorafenib which promoted tumor metastasis, and obviously prolong survival of a tumor-burdened nude mice.

So, the study is to observe the effect of sorafenib combined with aspirin in preventing the recurrence in high-risk patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The characteristics of the treatment history:

  1. No sorafenib treatment history, no sorafenib allergies.
  2. No chemotherapy, radiotherapy and transcatheter arterial chemoembolization(TACE) treatment history before surgery.
* The characteristics of the tumor:

  1. The pathological results is hepatocellular carcinoma.
  2. Meet any of the following articles:

     * Pathological prompt microvascular invasion(MVI) class II, and incorporate any of the following:Tumor number>3,Tumor size>8cm,Tumor margin is not clear and no complete capsule.
     * With the embolus in Portal vein, hepatic vein or bile duct.
     * Preoperative rupture or invasion the adjacent organs.
     * The positive cut edge.
     * Residual lesions showed by Postoperative digital subtraction angiography(DSA).
     * Alpha fetoprotein(AFP) did not drop to normal range two months after surgery.
* The characteristics of the patients:

  1. The patient age was between 18-75.
  2. The American Society of Anesthesiologists(ASA）score was I-III.
  3. No history of esophageal varices and gastrointestinal bleeding.
  4. The Child-pugh score was A.
  5. Routine blood test: the leukocyte>2.5*10^9, platelet> 60*10^9.
  6. The Prothrombin time was prolonged less than 2 second.
  7. The Eastern Cooperative Oncology Group(ECOG) score was less than 2 points

Exclusion Criteria:

* Sorafenib treatment before surgery.
* Pregnant or lactating women.
* The Child-pugh score was B-C.
* Patients with other malignant tumor.
* Patients with mental illness.
* Patients participated in other clinical trials in last three months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-04; Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years

SECONDARY OUTCOMES:
Disease free survival | 5 years
Number of patients with treatment-related bleedings who use aspirin | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lunxiu Qin, MD, Principal Investigator — Department of general surgery, Huashan hospital, Fudan University
Locations (1):
- Huashan hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Llovet JM, Burroughs A, Bruix J. Hepatocellular carcinoma. Lancet. 2003 Dec 6;362(9399):1907-17. doi: 10.1016/S0140-6736(03)14964-1. PMID 14667750
- [Result] Sun HC, Tang ZY, Wang L, Qin LX, Ma ZC, Ye QH, Zhang BH, Qian YB, Wu ZQ, Fan J, Zhou XD, Zhou J, Qiu SJ, Shen YF. Postoperative interferon alpha treatment postponed recurrence and improved overall survival in patients after curative resection of HBV-related hepatocellular carcinoma: a randomized clinical trial. J Cancer Res Clin Oncol. 2006 Jul;132(7):458-65. doi: 10.1007/s00432-006-0091-y. Epub 2006 Mar 24. PMID 16557381
- [Result] Llovet JM, Di Bisceglie AM, Bruix J, Kramer BS, Lencioni R, Zhu AX, Sherman M, Schwartz M, Lotze M, Talwalkar J, Gores GJ; Panel of Experts in HCC-Design Clinical Trials. Design and endpoints of clinical trials in hepatocellular carcinoma. J Natl Cancer Inst. 2008 May 21;100(10):698-711. doi: 10.1093/jnci/djn134. Epub 2008 May 13. PMID 18477802
- [Result] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Result] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Result] De Simone P, Crocetti L, Pezzati D, Bargellini I, Ghinolfi D, Carrai P, Leonardi G, Della Pina C, Cioni D, Pollina L, Campani D, Bartolozzi C, Lencioni R, Filipponi F. Efficacy and safety of combination therapy with everolimus and sorafenib for recurrence of hepatocellular carcinoma after liver transplantation. Transplant Proc. 2014 Jan-Feb;46(1):241-4. doi: 10.1016/j.transproceed.2013.10.035. PMID 24507059
- [Result] Bruix J, Takayama T, Mazzaferro V, Chau GY, Yang J, Kudo M, Cai J, Poon RT, Han KH, Tak WY, Lee HC, Song T, Roayaie S, Bolondi L, Lee KS, Makuuchi M, Souza F, Berre MA, Meinhardt G, Llovet JM; STORM investigators. Adjuvant sorafenib for hepatocellular carcinoma after resection or ablation (STORM): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2015 Oct;16(13):1344-54. doi: 10.1016/S1470-2045(15)00198-9. Epub 2015 Sep 8. PMID 26361969
- [Result] Gasic GJ, Gasic TB, Stewart CC. Antimetastatic effects associated with platelet reduction. Proc Natl Acad Sci U S A. 1968 Sep;61(1):46-52. doi: 10.1073/pnas.61.1.46. No abstract available. PMID 5246932
- [Result] Gasic GJ, Gasic TB, Murphy S. Anti-metastatic effect of aspirin. Lancet. 1972 Oct 28;2(7783):932-3. doi: 10.1016/s0140-6736(72)92581-0. No abstract available. PMID 4116642
- [Result] Rothwell PM, Wilson M, Elwin CE, Norrving B, Algra A, Warlow CP, Meade TW. Long-term effect of aspirin on colorectal cancer incidence and mortality: 20-year follow-up of five randomised trials. Lancet. 2010 Nov 20;376(9754):1741-50. doi: 10.1016/S0140-6736(10)61543-7. Epub 2010 Oct 21. PMID 20970847
- [Result] Rothwell PM, Fowkes FG, Belch JF, Ogawa H, Warlow CP, Meade TW. Effect of daily aspirin on long-term risk of death due to cancer: analysis of individual patient data from randomised trials. Lancet. 2011 Jan 1;377(9759):31-41. doi: 10.1016/S0140-6736(10)62110-1. Epub 2010 Dec 6. PMID 21144578
- [Result] Mahdi JG, Alkarrawi MA, Mahdi AJ, Bowen ID, Humam D. Calcium salicylate-mediated apoptosis in human HT-1080 fibrosarcoma cells. Cell Prolif. 2006 Aug;39(4):249-60. doi: 10.1111/j.1365-2184.2006.00390.x. PMID 16872361
- [Result] Saad-Hossne R, Prado RG, Hossne WS. Effects of acetylsalicylic acid and acetic acid solutions on VX2 liver carcinoma in rabbits. In vivo analysis. Acta Cir Bras. 2007 Jul-Aug;22(4):299-308. doi: 10.1590/s0102-86502007000400012. PMID 17625669
- [Result] Abiru S, Nakao K, Ichikawa T, Migita K, Shigeno M, Sakamoto M, Ishikawa H, Hamasaki K, Nakata K, Eguchi K. Aspirin and NS-398 inhibit hepatocyte growth factor-induced invasiveness of human hepatoma cells. Hepatology. 2002 May;35(5):1117-24. doi: 10.1053/jhep.2002.32676. PMID 11981761
- [Result] Zhang W, Sun HC, Wang WQ, Zhang QB, Zhuang PY, Xiong YQ, Zhu XD, Xu HX, Kong LQ, Wu WZ, Wang L, Song TQ, Li Q, Tang ZY. Sorafenib down-regulates expression of HTATIP2 to promote invasiveness and metastasis of orthotopic hepatocellular carcinoma tumors in mice. Gastroenterology. 2012 Dec;143(6):1641-1649.e5. doi: 10.1053/j.gastro.2012.08.032. Epub 2012 Aug 23. PMID 22922424
- [Result] Lu L, Sun HC, Zhang W, Chai ZT, Zhu XD, Kong LQ, Wang WQ, Zhang KZ, Zhang YY, Zhang QB, Ao JY, Li JQ, Wang L, Wu WZ, Tang ZY. Aspirin minimized the pro-metastasis effect of sorafenib and improved survival by up-regulating HTATIP2 in hepatocellular carcinoma. PLoS One. 2013 May 31;8(5):e65023. doi: 10.1371/journal.pone.0065023. Print 2013. PMID 23741443